CLINICAL TRIAL: NCT01471769
Title: Video Education Intervention in the Emergency Department
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, Amy Drendel, Principal Investigator: Assistant Professor, DO, MS, Medical College of Wisconsin
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: CHW 10/156
Record Dates: First submitted 2011-07-20; First posted 2011-11-16 (Estimated); Last update posted 2012-12-19 (Estimated); Status verified 2012-12

CONDITIONS: Pain
Keywords: pediatric; pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- pain management video (Experimental): Experimental
  Interventions: Behavioral: Pain management video
- falls prevention video (Placebo Comparator): placebo
  Interventions: Behavioral: Falls Prevention Video

INTERVENTIONS:
Behavioral: Pain management video — 6-minute video
  Arms: pain management video
Behavioral: Falls Prevention Video — 6-minute video
  Other Names: Fall Prevention Video
  Arms: falls prevention video

SUMMARY:
The purpose of this study is to evaluate if an educational video viewed during the Emergency Department visit will improve parent knowledge of pain management, reduce parent anxiety, and change their use of analgesics at-home after discharge from the Emergency Department.

DETAILED DESCRIPTION:
This study will investigate the use of a video instruction for parents just prior to discharge on pain treatment for their child. The investigators plan to investigate the effect of the video on knowledge because educational modules in the form of videotapes have been shown to be an effective method to improve a parent's knowledge about pain management prior to surgical procedures. Because parental anxiety has a significant impact on a child's experience of pain and video education has been shown to reduce parent anxiety before a procedure, the investigators will also evaluate if parental anxiety is reduced. Whether or not a short video will change the behavior of parents or their satisfaction with the outcome at home has not been investigated and will be an exploratory hypothesis for this study. This research will be a first step towards optimizing the outpatient care for common diagnoses in the Emergency Department.

ELIGIBILITY:
Inclusion Criteria:

* complaint of pain or injury and laceration, fracture or spring, contusion, crush injuries, head injury, motor vehicle collision, or burn.

Exclusion Criteria:

* non- English speaking parents
* primary caregiver not with child in Emergency Department

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Actual)
Dates: Start 2011-06; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Change in parent knowledge from baseline | on day 0 in the ED
  A parent knowledge test will be completed by parents prior to the video intervention, immediately after the video intervention, and on day 3 after the video intervention.

SECONDARY OUTCOMES:
Change in anxiety from baseline | on day 0 in the ED
  Parent's anxiety will be measured using a validated pain scale before and immediately after the video intervention
Pain medication use | assessed on day 0, 1, 2, 3
  Pain medicatin use collected in a diary at-home after ED treatment
Child's pain | on day 0, 1, 2, 3
  child's reported pain at-home after ED treatment
satisfaction | on day 1, 2, and 3
  child and parent at-home satisfaction utilizing a validated likert scale will be assesed on day 1, 2, and 3 after ED treatment to determine if the intervention results in improved satisfaction with pain treatment after discharge home

CONTACTS AND LOCATIONS:
Overall Officials: Amy L Drendel, DO, Principal Investigator — Medical College of Wisconsin
Locations (1):
- Children's Hospital of Wisconsin, Milwaukee, Wisconsin, United States